CLINICAL TRIAL: NCT00179192
Title: Prevention and Treatment of Hemodialysis Vascular Access Malfunction
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: non-enrollment
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Alp Ikizler, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9318
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: End-Stage Renal Disease
Keywords: End Stage Renal Disease; ESRD; Chronic Maintenance Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Angioplasty; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): control group
- 2 (Active Comparator): angioplasty intervention
  Interventions: Procedure: angioplasty
- 3 (Active Comparator): surgery intervention
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: angioplasty — angioplasty performed at the time of the angiogram; approach and technique to be determined by the interventional radiologist
  Arms: 2
Procedure: surgery — surgical revision of patient's PTFE in a timely fashion not to exceed 72-96 hours after the angiogram; method of revision to be determined by the surgeon performing the procedure
  Arms: 3

SUMMARY:
Vascular access is considered the Achilles heel of the dialysis patient. It constitutes the largest single cause of morbidity in the chronic hemodialysis population, accounting for over 25% of hospitalizations at an estimated cost in the US of at least one billion dollars annually. Currently, complication free survival of vascular access ranges between 30-50% a year and multiple investigative efforts in this area have been initiated and are directed at prolonging the functional life of vascular accesses.

It is not well established whether intervention prior to overt malfunction or thrombosis of the vascular access could reduce these complications and thereby improve the functional longevity of the access. Moreover, once accesses at potential risk are identified, it is not well established which method of intervention, Surgery vs. Angioplasty vs. Expectant Management, is superior in terms of clinical and financial outcome. The proposed study aims to determine whether early intervention of a vascular access determined to be at risk of malfunction and thrombosis improves the long term outcome and, specifically, which means of intervention is preferred.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with End Stage Renal Disease on chronic maintenance hemodialysis 3 times per week
2. Have an arteriovenous (polytetrafluoroethylene) graft as vascular access
3. Have a venous stenosis between 30% and 70% as determined by angiogram

Exclusion Criteria:

1. Native arteriovenous fistula
2. Known previous vascular accesses complications, such as central vein stenosis, and multiple access surgeries >4
3. Unwilling to participate
4. Allergy to iodine
5. Absolute contraindication for surgery (e.g. medical condition precludes anesthesia and surgery)
6. Known arterial limb stenosis or long vessel length venous stenosis which are unamenable to surgical or angioplasty techniques, respectively, and therefore prohibit randomization
7. Known hypercoagulable state

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1998-05; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
To test the hypothesis that early intervention of a vascular access determined to be at increased risk of malfunction and thrombosis improves the long-term access outcome versus standard of care. | 2 years

SECONDARY OUTCOMES:
To determine which means of early intervention, surgery versus angioplasty, is medically and financially advantageous. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Talat A Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States